CLINICAL TRIAL: NCT05847738
Title: Comparative Evaluation of Post-operative Pain With Different Apical Finishing Sizes After Single Visit Root Canal Treatment
Brief Title: Post-operative Pain With Different Apical Finishing Sizes After Single Visit Root Canal Treatment
Status: Completed | Type: Observational
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Hala Fayek, Associate Professor, British University In Egypt
Other Study IDs: FD-BUE-REC 23-002
Record Dates: First submitted 2023-04-19; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Pain Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: (left side of the patient: prepared 2 sizes larger than the IBF, to size 35#/.04 mesial canals and 40#/.04 distal canals.
  Interventions: Behavioral: Pain assessment
- Group B (right side of the patient: prepared 3 sizes larger than the IBF, to size 40#/.04 mesial canals and 45#/.04 distal canals.
  Interventions: Behavioral: Pain assessment

INTERVENTIONS:
Behavioral: Pain assessment — Pain was assesd postoperatively in both groups at time intervals

SUMMARY:
This is a randomized controlled parallel clinical, prospective split mouth, triple blinded study. Sample size calculation was conducted and it was 25 subjects per group for a total of 50 sides to compensate for drop-outs.

Patient selection and preparation:

All root canal treatments were performed by a single endodontic consultant. All subjects were selected from walk in patients presented to the endodontic clinic of the British university in Egypt. Cases that met the inclusion criteria where selected for this study. All patients were verbally informed about the procedure's benefits and that the results of the treatment will be used to this study and the risks of the procedure was explicitly explained to them. After the verbal consent patients were handed a written form consent to sign upon.

All data of post-operative pain were recorded by a second blinded clinician through a visual analog scale (VAS). Post-operative monitoring periods will be recorded in 12 hours, 24 hours, 3 days and one week Data was sent to the statistician with group names only to fulfill the triple blinding criteria and results will be interpreted

DETAILED DESCRIPTION:
This is a randomized controlled parallel clinical, prospective split mouth, triple blinded study. Sample size calculation was conducted using G*Power 3.1.9.4 software based on data obtained from a previous study ] It was estimated that a minimum sample size of 19 subjects (sides) per group for a total of 38 sides would be essential for an effect size of 0.97 with an alpha error of 0.05 and a power beta of 0.90 to achieve 95% confidence of a true difference between the groups. Sample size was increased by 25% to 25 subjects per group for a total of 50 sides to compensate for drop-outs.

Patient selection and preparation:

All root canal treatments were performed by a single endodontic consultant. All subjects were selected from walk in patients presented to the endodontic clinic of the British university in Egypt. Cases that were diagnosed and did not meet the inclusion criteria were referred to the intern clinic for dental care. Cases that met the inclusion criteria where selected for this study. All patients were verbally informed about the procedure's benefits and that the results of the treatment will be used to this study and the risks of the procedure was explicitly explained to them. After the verbal consent patients were handed a written form consent to sign upon.

Procedure:

Radiographs were taken by a Paralleled long cone periapical radiography. To ensure a visible root canal ≤30° of canal curvature and a periapical index (PAI score) of 3-5 in addition of initial confirmation of root canal types. All patients were anesthetized, rubber dam applied, and access cavities were performed. After root canal exploration and scouting, root canal systems were reconfirmed to be the types selected for this study.

Initial binding file was selected for all root canals to ensure it met the inclusion size of mesial roots #20 and distal #30. After patency and glide path were performed by K-files up to size #20, engine driven canal enlargement was applied using E3 Azure files to final finishing size according to the grouping.

Group A: (left side of the patient) were prepared 2 sizes larger than the IBF, to size 35#/.04 mesial canals and 40#/.04 distal canals.

Group B: (right side of the patient) were prepared 3 sizes larger than the IBF, to size 40#/.04 mesial canals and 45#/.04 distal canals.

All data of post-operative pain were recorded by a second blinded clinician through a visual analog scale (VAS). Post-operative monitoring periods will be recorded in 12 hours, 24 hours, 3 days and 1 week.

Data was sent to the statistician with group names only to fulfill the triple blinding criteria and results will be interpreted

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50
* Gender: Males and Females, random selection.
* Systemic status: healthy patients (Category: American Society of Anaesthesiologists class 1)
* Bilateral exposed mandibular first or second permanent molars
* Molars should have separate mesial and distal roots
* Mesial roots confirmed to be type three root canal system
* Distal root confirmed to be type one root canal system
* Normal periapical radiograph and no bone changes
* Symptomatic irreversible pulpitis
* I.B.F. in mesial roots not more than #20, and distal root not more than #30

Exclusion Criteria:

* Type two root canal system in mesial roots
* Type two or three root canal systems in distal roots
* Signs of apical involvement in the radiograph
* Any systemic conditions altering the treatment or requiring medications or precautions

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All types of adult population
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Pain assessment at 12 hours | 12 hours
  post-operative pain will be recorded by a second blinded clinician using a visual analog scale where patient grades his level of pain from minimum to maximum Post-operative monitoring periods wiere recorded
Pain assessment at 24 hours | 24 hours
  Comparative post-operative pain will be recorded by a second blinded clinician using a visual analog scale where patient grades his level of pain from minimum to maximum Post-operative monitoring periods wiere recorded
Pain assessment at 3 days | 3days
  post-operative pain will be recorded by a second blinded clinician using a visual analog scale where patient grades his level of pain from minimum to maximum Post-operative monitoring periods wiere recorded
Pain assessment at 1 week | 1 week
  post-operative pain will be recorded by a second blinded clinician using a visual analog scale where patient grades his level of pain from minimum to maximum Post-operative monitoring periods wiere recorded

CONTACTS AND LOCATIONS:
Locations (1):
- British university, Cairo, El Shrouk, Egypt

REFERENCES:
- [Derived] Kataia MM, Kataia EM, Khalil HF, Seoud MAE. Post-operative pain after root canal preparation with different apical finishing sizes a triple blinded split mouth clinical trial. BMC Oral Health. 2024 Jul 16;24(1):800. doi: 10.1186/s12903-024-04527-9. PMID 39014316

DOCUMENTS (1):
  • Study Protocol (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT05847738/Prot_000.pdf